CLINICAL TRIAL: NCT06383078
Title: HR070803 in Combination With Oxaliplatin Plus Tegafur Versus HR070803 in Combination With Oxaliplatin, 5-fluorouracil, Calcium Folinate as Adjuvant Therapy for Pancreatic Cancer: A Multicenter, Multi-cohort, Randomized, Phase II Study
Brief Title: HR070803 in Combination With Oxaliplatin, S-1 Versus NALIRIFOX as Adjuvant Therapy for Pancreatic Cancer
Status: Not yet recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: The First Affiliated Hospital with Nanjing Medical University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MA-PC-II-012
Record Dates: First submitted 2024-04-03; First posted 2024-04-25 (Actual); Last update posted 2024-04-25 (Actual); Status verified 2024-04

CONDITIONS: Efficacy and Safety
MeSH Terms: interventions — irinotecan sucrosofate; Oxaliplatin; Tegafur; S 1 (combination); Leucovorin; Fluorouracil

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HR070803+Oxaliplatin+S-1 (Experimental): Drug: HR070803（Irinotecan Liposome）; Oxaliplatin; Tegafur HR070803 60 mg/^2 D1 over 90 minutes. Oxaliplatin 85 mg/^2 D1 over 2 hours. Tegafur The initial dose of S-1 is determined according to the body surface area，orally, D1-7.
  These drugs are given once every 2 weeks, 4 weeks as one cycle, 6 treatment cycles.
  Interventions: Drug: HR070803; Drug: Oxaliplatin; Drug: Tegafur
- HR070803+Oxaliplatin+5-FU/LV (Active Comparator): Drug: HR070803; Oxaliplatin; 5-Fluorouracil; Calcium folinate HR070803 60 mg/^2 D1 over 90 minutes. Oxaliplatin 85 mg/^2 D1 over 2 hours. Folinic acid 400 mg/^2 D1, IV infusion over 1 hours. 5-FU 2400 mg/^2 D1 IV continuous infusion over 46 hours.
  These drugs are given once every 2 weeks, 4 weeks as one cycle, 6 treatment cycles.
  Interventions: Drug: HR070803; Drug: Oxaliplatin; Drug: Folinic acid; Drug: 5-Fluorouracil

INTERVENTIONS:
Drug: HR070803 — HR070803 60 mg/^2 D1 over 90 minutes.
  Other Names: Irinotecan Liposome
Drug: Oxaliplatin — Oxaliplatin 85 mg/^2 D1 over 2 hours.
  Other Names: L-OHP
Drug: Tegafur — initial dose of S-1 is determined according to the body surface area，orally, D1-7.
  Other Names: S-1
  Arms: HR070803+Oxaliplatin+S-1
Drug: Folinic acid — Folinic acid 400 mg/^2 D1
  Other Names: LV
  Arms: HR070803+Oxaliplatin+5-FU/LV
Drug: 5-Fluorouracil — 5-FU 2400 mg/^2 D1 IV continuous infusion over 46 hours
  Other Names: 5-FU
  Arms: HR070803+Oxaliplatin+5-FU/LV

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of HR070803 in Combination With Oxaliplatin plus Tegafur compared to HR070803 in combination with oxaliplatin, 5-fluorouracil/leucovorin (5FU/LV) treatment as adjuvant therapy in patients with resected pancreatic cancer.

DETAILED DESCRIPTION:
STUDY DESIGN/ Evaluation criteria Main criterion: efficacy. The main criterion is the 1-year disease-free survival rate. Disease-free survival is defined as the time from date of randomization until the date of the first cancer-related event, second cancer, or death from any cause. Patients without event at the time of analysis will be censored at the date of last follow-up visit.

Secondary criteria include Overall survival. OS is defined as the time from date of randomization until the date of death from any cause. Patients who are still living at the time of analysis will be censored at the date of last follow-up visit.

Secondary criteria also include the Disease-free survival.

Tolerance Patients evaluable for toxicity must have received one investigational drug.

ELIGIBILITY:
Inclusion Criteria:

1. Histologically confirmed resected ductal pancreatic adenocarcinoma with macroscopic complete resection (R0 and R1).
2. ECOG performance status 0 or 1.
3. Life expectancy of greater than or equal to 6 months.
4. Full recovery from surgery and patient is scheduled to start treatment within 3 weeks to 12 weeks after surgery.
5. The number of lymph nodes dissected during resection ≥ 15.
6. Able and willing to provide a written informed consent.

Exclusion Criteria:

1. Patients with pancreatic cancer originating from extrapancreatic ductal epithelium, including pancreatic neuroendocrine carcinoma, acinar cell carcinoma of the pancreas, pancreatoblastoma, and solid-pseudopapillary tumor;
2. Presence of or history of metastatic or locally recurrent pancreatic adenocarcinoma.
3. CA19-9 exceeding normal value within 14 days prior to enrollment.
4. Prior neo-adjuvant treatment, radiation therapy, or systemic therapy for pancreatic adenocarcinoma.
5. Severe infection (> CTCAE grade 2), such as severe pneumonia, bacteremia, infection complications, etc. requiring inpatient treatment, occurred within four weeks before enrollment, and symptoms and signs of infection requiring intravenous antibiotic therapy (except for prophylactic antibiotics) occurred within two weeks before enrollment;
6. Patients with cardiac clinical symptoms or diseases that are not well controlled, such as: (1) Patients with NYHA class 2 and above cardiac failure; (2) unstable angina; (3) myocardial infarction that occurred within 6 months; (4) clinically significant supraventricular or ventricular arrhythmia requiring treatment or intervention.

Ages: 20 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2024-04-20 (Estimated); Primary Completion 2027-03-01 (Estimated); Study Completion 2027-12-30 (Estimated)

PRIMARY OUTCOMES:
1-year Disease-free survival rate | Up to 2 years
  Disease-free survival is defined as the time from date of randomization until the date of the first cancer-related event, second cancer, or death from any cause.

SECONDARY OUTCOMES:
Overall survival (OS) | Up to 2 years
  OS is defined as the time from date of randomization until the date of death from any cause.
Disease-free survival（DFS） | Up to 2 years
  Disease-free survival is defined as the time from date of randomization until the date of the first cancer-related event, second cancer, or death from any cause.

IPD SHARING:
Plan to Share IPD: No
There is not a plan to make individual participant data (IPD) available to other researchers.